CLINICAL TRIAL: NCT04253834
Title: GO2 PEEP Study: The Use of a Bidirectional Oxygenation Valve in the Prevention and Management of Postoperative Atelectasis
Brief Title: GO2 PEEP Study: Bidirectional Oxygenation Valve in Postoperative Atelectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: PEEP Medical, LLC (Industry)
Responsible Party: Principal Investigator, Jeffrey Miller, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00117254
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Atelectasis
Keywords: Cardiac surgery; Coronary bypass; Heart valve replacement; Postoperative pulmonary complications

STUDY DESIGN:
Intervention Model Description: Single center, prospective, randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Incentive Spirometer Control Arm (Active Comparator): Participants assigned to use the incentive spirometer after surgery.
  Interventions: Device: Incentive spirometer
- GO2 Mouthpiece (Experimental): Participants assigned to use the Bidirectional Oxygenation Valve (GO2 Mouthpiece) after surgery.
  Interventions: Device: GO2 Mouthpiece

INTERVENTIONS:
Device: Incentive spirometer — The incentive spirometer is a device that measures how deeply a person can inhale (breathe in). It helps with taking slow, deep breaths to expand and fill the lungs with air, which helps prevent lung problems, such as pneumonia. The incentive spirometer is made up of a breathing tube, an air chamber, and an indicator to help users control their breathing.
  Arms: Incentive Spirometer Control Arm
Device: GO2 Mouthpiece — The GO2 Mouthpiece is a simple, comfortable, and straightforward silicone rubber-made, bidirectional oxygenation mouthpiece that effectively delivers PEEP with every breath.
  Other Names: Bidirectional Oxygenation Valve
  Arms: GO2 Mouthpiece

SUMMARY:
This study compares a novel breathing device, called the GO2 Mouthpiece, to the standard breathing tool called the incentive spirometer, thus improving respiratory dynamics of the postoperative patient.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) are the principal cause of morbidity, mortality and prolonged hospitalizations in surgical patients, which results in a 50% increase in healthcare costs compared to postoperative cardiac complications. This is especially evident following cardiovascular surgery. One of the most common PPCs is atelectasis, resulting in dyspnea, tachypnea and hypoxemia.

Postoperative atelectasis is a predictable consequence of anesthesia, surgical trauma, and pain associated with breathing. Methods aimed at increasing lung volume and treating atelectasis, commonly known as postoperative physiotherapy, play an important role in preventing PPCs. These methods include cough and deep breathing, continuous positive airway pressure (CPAP), postural drainage, incentive spirometry and positive end expiratory pressure (PEEP).

Incentive spirometry has served as a convenient approach for the postoperative patient to sustain maximal inflations and encourage deep breathing. Although incentive spirometry is used commonly by post-operative patients, evidence fails to support its benefit.

PEEP is a well-known pulmonary physiologic principle. There are on average 600 million alveoli in the lung. Each alveolus has surfactant to resist the natural propensity for these small air sacs to collapse during exhalation. Despite this surfactant, some alveoli will collapse and not be available for gas exchange. This atelectasis results in a ventilation/perfusion mismatch where alveolar units are perfused but not adequately ventilated. This is referred to as shunting and results in hypoxemia (decreased PaO2). PEEP decreases the propensity for the alveoli to collapse by increasing the air pressure in the lungs. This residual pressure in the lungs at the end of exhalation decreases shunting and allows for more complete gas exchange and improved oxygenation. In patients, PEEP is one of the safest ways to increase PaO2 and is used on almost all modern ventilator settings.

The purpose of this study is to compare a novel breathing device, called the GO2 Mouthpiece, which uses the concept of PEEP, to the incentive spirometer in postoperative patients.

ELIGIBILITY:
Inclusion Criteria

1. Undergoing coronary artery bypass surgery (CABG) and/or valve replacement surgery
2. Able to provide written informed consent
3. Maintenance of an arterial line postoperatively

Exclusion Criteria

1. Active smoking, within three months of surgery
2. Forced expiratory volume in one second (FEV1) <75% predicted
3. Relative risk to develop pulmonary barotrauma as evident by history of pneumothorax or emphysema
4. Unable or unwilling to provide informed consent, cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Emory University
Locations (1):
- Emory Saint Joseph's Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began August 27, 2020 and all study follow up was completed January 31, 2021. Participants were enrolled at Emory Saint Joseph's Hospital in Atlanta, Georgia, USA.
Groups:
- Incentive Spirometer Control Arm: Participants using the incentive spirometer after surgery.
- GO2 Mouthpiece: Participants using the bidirectional oxygenation valve, GO2 Mouthpiece, after surgery.
Period: Overall Study
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GO2 Mouthpiece: Participants using the GO2 Mouthpiece after surgery.
- Total: Total of all reporting groups
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.7) | 67.1 (6.9) | 66.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Partial Pressure of Oxygen (PaO2 Level)
Description: Partial pressure of oxygen is a measurement of oxygen pressure in arterial blood. It reflects how well oxygen is able to move from the lungs to the blood. Normal values are 80 to 100 millimeters of mercury (mmHg).
Time Frame: 1, 6, 12 and 24 hours postextubation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
mmHg
  1 hour postextubation | 95.4 (22.6) | 83.5 (18.3)
  6 hours postextubation | 92.1 (28.1) | 85.4 (22.3)
  12 hours postextubation | 91.0 (21.8) | 81.4 (17.9)
  24 hours postextubation | 74.5 (17.2) | 77.8 (14.6)

2. Secondary Outcome: Number of Participants With Normal Atelectasis Score
Description: Atelectasis is a lung condition that happens when the airways don't expand normally. Atelectasis is measured with the modified radiological atelectasis score (m-RAS). Each pulmonary lobe, including the lingula, is scored 0-3 (0=normal, 1=plate or minor infiltrate, 2= moderate atelectasis, 3= total atelectasis). The scores of the six lobes are then summed to give a total score ranging from 0 to 18 with higher scores being associated with worse outcomes. For this analysis, scores were categorized as 0 (normal) or greater than 0 (not normal). The count of participants with a normal atelectasis score at the indicated time point are presented here.
Time Frame: Immediately postoperative, Postoperative days 1, 2, 3, 4
Population: This analysis includes participants who completed the chest x-ray at the indicated visits. The atelectasis score could not be determined for one participant at postoperative day 3 and two participants at postoperative day 4 because chest x-rays were not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
Participants
  Immediately Postoperative | 0 | 2
  Postoperative Day 1 | 0 | 0
  Postoperative Day 2 | 0 | 0
  Postoperative Day 3: number analyzed (Participants) | 9 | 10
  Postoperative Day 3 | 0 | 0
  Postoperative Day 4: number analyzed (Participants) | 9 | 9
  Postoperative Day 4 | 2 | 0

3. Secondary Outcome: Oxygen Requirement
Description: Oxygen was provided by a nasal cannula. The flow rate of supplemental oxygen that participants required after surgery is assessed as liters per minute. Higher flow rate indicates an increased need for supplemental oxygen.
Time Frame: Postextubation Hours 1, 6, 12 and 24, Postoperative Days 2, 3, and 4
Measure: Mean (Standard Deviation); unit: liters of oxygen per minute
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
liters of oxygen per minute
  Postextubation Hour 1 | 3.7 (1.26) | 3.7 (1.7)
  Postextubation Hour 6 | 2.3 (0.7) | 2.4 (0.8)
  Postextubation Hour 12 | 2.2 (1.5) | 2.1 (0.3)
  Postextubation Hour 24 | 2.4 (2.8) | 2.3 (0.7)
  Postoperative Day 2 | 2.0 (1.6) | 2.3 (1.1)
  Postoperative Day 3 | 1.1 (1.2) | 1.7 (0.9)
  Postoperative Day 4 | 0.6 (1.0) | 0.5 (1.1)

4. Secondary Outcome: Carbon Dioxide Level
Description: Normal carbon dioxide (CO2) levels in blood range from 35.0 mmHg to 45.0 mmHg.
Time Frame: Postextubation Hours 1, 6, 12 and 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
mmHg
  Postextubation Hour 1 | 38.2 (2.9) | 39 (3.3)
  Postextubation Hour 6 | 37.0 (4.8) | 37.2 (4.4)
  Postextubation Hour 12 | 37.3 (5.1) | 36.9 (4.2)
  Postextubation Hour 24 | 36.8 (5.1) | 38.1 (3.8)

5. Secondary Outcome: FEV1
Description: Forced expiratory volume in one second (FEV1) is measured during a spirometry test, also known as a pulmonary function test, which involves forcefully breathing out into a mouthpiece connected to a spirometer machine.
  FEV1 is the amount of air forced from lungs in one second. To describe severity of pulmonary disease, FEV1 can be expressed as a percentage of the predicted value. Values 80% and and greater of the predicted value are considered normal.
Time Frame: Preoperative and postoperative day 3
Measure: Mean (Standard Deviation); unit: percentage of the predicted FEV1 value
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
percentage of the predicted FEV1 value
  Preoperative | 86.4 (10.1) | 93.7 (8.9)
  Postoperative Day 3 | 35.9 (8.0) | 43.1 (10.7)

6. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is measured during a spirometry test, also known as a pulmonary function test, which involves forcefully breathing out into a mouthpiece connected to a spirometer machine. FVC is the total amount of air exhaled during the FEV test. FVC can be expressed as a percentage of the predicted value.The normal range for the percent of the predicted value is between 80% and 120%.
Time Frame: Preoperative, Postoperative Day 3
Measure: Mean (Standard Deviation); unit: percentage of the predicted FVC value
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
percentage of the predicted FVC value
  Preoperative | 85.7 (9.8) | 90.1 (8.3)
  Postoperative Day 3 | 38.0 (9.9) | 41.6 (10.5)

7. Secondary Outcome: Respiratory Rate
Description: Respiratory rate is the number of breaths taken per minute. The normal respiration rate for an adult at rest is 16 to 20 breaths per minute.
Time Frame: Postextubation Hours 1, 6, 12 and 24, Postoperative Days 2, 3, and 4
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
breaths per minute
  Postextubation Hour 1 | 21.3 (4.0) | 20.5 (5.8)
  Postextubation Hour 6 | 21.2 (5.5) | 17.9 (4.8)
  Postextubation Hour 12 | 21.0 (3.9) | 19.2 (3.3)
  Postextubation Hour 24 | 20.7 (3.8) | 18.9 (3.2)
  Postoperative Day 2 | 21.7 (4.9) | 20.6 (3.4)
  Postoperative Day 3 | 18.4 (1.3) | 18.4 (1.3)
  Postoperative Day 4 | 18.0 (1.7) | 18.6 (1.3)

8. Secondary Outcome: Body Temperature
Description: Measure of heat associated with the metabolism of the body. Normal range is between 36.5-37.5 degrees Celsius (°C).
Time Frame: Immediately Postoperative, Postoperative Day 1, 2, 3, 4
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Incentive Spirometer Control Arm | GO2 Mouthpiece
Number analyzed (Participants) | 10 | 10
°C
  Postoperative | 36.8 (0.2) | 36.8 (0.3)
  Postoperative Day 1 | 38.0 (1.4) | 37.7 (0.4)
  Postoperative Day 2 | 37.5 (0.4) | 37.4 (0.3)
  Postoperative Day 3 | 37.3 (0.3) | 37.4 (0.3)
  Postoperative Day 4 | 37.2 (0.2) | 37.2 (0.2)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the initial postoperative assessment and was collected through postoperative day 4.
Groups:
- Control Arm: Participants using the incentive spirometer after surgery.
Arm/Group | Control Arm | GO2 Mouthpiece
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=10) | GO2 Mouthpiece (N=10)
Increased oxygen requirement 10% (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Bilevel positive airway pressure (BiPAP) requirement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT04253834/Prot_SAP_000.pdf